CLINICAL TRIAL: NCT02694432
Title: An Internet-Assisted Mind-Body-Behavior Program for Blood Pressure Control
Brief Title: Minding GOALS: An Internet-Assisted Mind-Body-Behavior Program for Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Natalia Morone, Associate Professor of Medicine & Clinical and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO15120045; R34HL123500-01 (NIH)
Record Dates: First submitted 2016-01-12; First posted 2016-02-29 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: high blood pressure, systolic, diastolic; complementary therapies, meditation
MeSH Terms: conditions — Hypertension; Systolic Murmurs; Heart Murmurs | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GOALS (Active Comparator): Participants will use for approximately four months an online platform, GOALS, consisting of weekly lessons designed to enhance blood pressure control. Recommended lifestyle changes for hypertension, including a low-sodium diet, physical activity, weight loss (if appropriate) and behavioral self-management skills will be offered. Attention to medication adherence and pharmacist support as well as that of a dedicated online health coach and ongoing collaboration with the primary care physician are also provided.
  Interventions: Behavioral: GOALS
- Minding GOALS (Experimental): Participants in this arm will also use the GOALS standard tools for blood pressure control. To further maximize success, they will receive additional online behavioral training throughout the 4-month intervention that focuses on mind-body approaches. Weekly topics, for example, will include meditation lessons, mindfulness-based stress reduction and mindfulness-based eating awareness.
  Interventions: Behavioral: GOALS; Behavioral: Minding GOALS

INTERVENTIONS:
Behavioral: GOALS — 16 weeks of online support to improve blood pressure using traditional behavioral lifestyle approaches and medication adherence support.
Behavioral: Minding GOALS — 16 weeks of online support to improve blood pressure using traditional behavioral lifestyle approaches and medication adherence support, coupled with a mind-body-behavior program to further enhance improvements in blood pressure.
  Other Names: Stress reduction
  Arms: Minding GOALS

SUMMARY:
This pilot study will evaluate the feasibility of adding an online mind-body-behavior program to an existing behavioral self-management support platform that has been modified to promote achievement of blood pressure goals.

DETAILED DESCRIPTION:
Efficacious hypertension therapies are well-documented, yet 40% of treated patients do not meet the blood pressure goals set by the Joint National Committee. This gap between scientific evidence and clinical outcomes in part reflects low patient adherence to lifestyle recommendations (e.g., physical activity, weight and diet), as well as medication non-adherence. Accordingly, growing attention is focused on the need to provide patients with effective self-management support tools. In addition to finding ways to help patients adhere to currently prescribed hypertension care, it is useful to consider the range of treatment options that are offered. Evidence-based reviews have identified stress reduction as an effective tool for reducing blood pressure, yet such approaches are typically not implemented in practice. This omission represents a chance to improve the quality of hypertension care by adding stress management self-management tools. Furthermore, since patients have demonstrated a clear interest in mindfulness, the incorporation of a holistic mind-body intervention is an innovative approach to inherently patient-centered care. Increasing data supports the use of mindfulness for treating health concerns. Its holistic nature may be particularly well-suited to developing and maintaining healthy lifestyles, since lifestyle impacts diverse aspects of physical and psychological health. Yet the potential for mindfulness in health self-management has not been realized.

Limited but promising data demonstrate the effectiveness of web-based counseling for behavior modification to improve common chronic disease risk factors. It is an ideal solution to provider time constraints and a potential solution to patient non-adherence to lifestyle recommendations. Health information technology provides a way to make self-management support affordable, convenient and feasible. The investigators have developed a convenient behavioral self-management support platform, "Goal-oriented Online Access to Lifestyle Support" (GOALS) for primary care patients, which has promoted weight loss and improved blood pressure control among primary care patients with weight-related cardiovascular risk factors. To maximize the ability of patients to achieve blood pressure goals, the investigators propose to add an online mind-body-behavior program to GOALS: "Minding GOALS." The investigators will evaluate the feasibility of using this program for self-management support, in coordination with primary care, in a group of 76 patients with uncontrolled hypertension. In preparation for a randomized clinical trial comparing the online tool to online traditional self-management support, the investigators will assess implementation and determine 1) the availability of eligible and willing subjects using the proposed recruitment methods, 2) the feasibility of delivering the proposed interventions in the population of interest, and 3) the viability of the proposed measurement protocols.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure >/= 150 mmHg and/or
* Diastolic blood pressure >/= 90 mmHg and
* At least one other cardiovascular disease (CVD) risk factor (i.e., diabetes, dyslipidemia, family history of premature CVD, current smoking, obesity)

Exclusion Criteria:

* Known secondary hypertension of any etiology, malignant hypertension or hypertensive encephalopathy
* Severe edema
* A primary care physician (PCP) of the opinion that the patient is unable to safely undertake moderately intense unsupervised physical activity (equivalent of 30 minutes brisk walking)
* A PCP of the opinion that the patient has inadequate cognitive function to participate
* Previous participation in a mindfulness meditation program
* An inability to learn adequately from English language materials
* Current pregnancy or planned pregnancy within the next year
* A prior diagnosis of post-traumatic stress disorder
* Prior use of GOALS

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-09; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure and diastolic blood pressure (mm Hg) | Baseline, 4- and 12-months
  Change in blood pressure

SECONDARY OUTCOMES:
Change in sodium excretion (mmol/24 hr.) | Baseline and 12-months
  From 24-hr urine collection
Body weight (kg) | Baseline, 4- and 12-months
Body Mass Index (kg/m2) | Baseline, 4- and 12-months
Physical activity (steps/day) | Baseline, 4- and 12-months
  Assessed by pedometer
Health-related quality of life | Baseline, 4- and 12-months
  PROMIS (Patient Reported Outcomes Measurement Information System)-29 Profile v2.0
Perceived Stress Scale | Baseline, 4- and 12-months
PROMIS-29 Profile v2.0 | Baseline, 4- and 12-months
  Quality of Life
Mindful Attention Awareness Scale | Baseline, 4- and 12-months
  Assesses a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present
Self-reported medication adherence questions | Baseline, 4- and 12-months
  Self-reported scale to measure medication adherence
Credibility/Expectancy Questionnaire | Baseline, 4- and 12-months
  For measuring treatment expectancy and rationale credibility in clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Morone, MD, MS, Principal Investigator — University of Pittsburgh; Kathleen M McTigue, MD, MS, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Center for Research on Health Care, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McTigue KM, Conroy MB, Hess R, Bryce CL, Fiorillo AB, Fischer GS, Milas NC, Simkin-Silverman LR. Using the internet to translate an evidence-based lifestyle intervention into practice. Telemed J E Health. 2009 Nov;15(9):851-8. doi: 10.1089/tmj.2009.0036. PMID 19919191
- [Background] McTigue KM, Bhargava T, Bryce CL, Conroy M, Fischer GS, Hess R, Simkin-Silverman LR, Zickmund S. Patient perspectives on the integration of an intensive online behavioral weight loss intervention into primary care. Patient Educ Couns. 2011 May;83(2):261-4. doi: 10.1016/j.pec.2010.05.009. Epub 2010 Jun 17. PMID 21459256
- [Background] McTigue KM, Conroy MB. Use of the internet in the treatment of obesity and prevention of type 2 diabetes in primary care. Proc Nutr Soc. 2013 Feb;72(1):98-108. doi: 10.1017/S0029665112002777. Epub 2012 Oct 26. PMID 23098133
- [Background] Morone NE, Greco CM, Weiner DK. Mindfulness meditation for the treatment of chronic low back pain in older adults: a randomized controlled pilot study. Pain. 2008 Feb;134(3):310-319. doi: 10.1016/j.pain.2007.04.038. Epub 2007 Jun 1. PMID 17544212
- [Background] Morone NE, Lynch CS, Greco CM, Tindle HA, Weiner DK. "I felt like a new person." the effects of mindfulness meditation on older adults with chronic pain: qualitative narrative analysis of diary entries. J Pain. 2008 Sep;9(9):841-8. doi: 10.1016/j.jpain.2008.04.003. Epub 2008 Jun 12. PMID 18550444
- [Background] Simkin-Silverman LR, Conroy MB, Bhargava T, McTigue KM. Development of an online diabetes prevention lifestyle intervention coaching protocol for use in primary care practice. Diabetes Educ. 2011 Mar-Apr;37(2):263-8. doi: 10.1177/0145721710396587. PMID 21421991
- [Background] Morone NE, Greco CM, Rollman BL, Moore CG, Lane B, Morrow L, Glynn NW, Delaney J, Albert SM, Weiner DK. The design and methods of the aging successfully with pain study. Contemp Clin Trials. 2012 Mar;33(2):417-25. doi: 10.1016/j.cct.2011.11.012. Epub 2011 Nov 15. PMID 22115971